CLINICAL TRIAL: NCT06672042
Title: Parental AdheRence of an Asynchronous Mobile hEalth Application for Children With Medical TEchnologies Using a Randomized Trial of Outpatient Nursing Care Models (PARAMETER)
Brief Title: Parental Adherence of a Mobile Application
Acronym: PARAMETER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been withdrawn/stopped as funding was not recieved. Therefore, study was never started (no participants enrolled).
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Lori Erickson, Director, Remote Health Solutions, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00003221
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pediatrics; Medically Complex; Children With Medical Complexity (CMC); Nursing
Keywords: mHealth; Software Platform; remote patient monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Proactive Nursing Care model using a mobile application and software platform (Experimental): * Includes weekly data monitoring by the study team clinical nurse coordinators with communication through phone, email, or patient portal with documentation in the EMR
  * Email delivery of data summary reports on each child's data to their outpatient providers, Unrestricted research team approved healthcare team provider access to this data through the CHAMP App PARAMETER web portal,
  * Follow-up communications from providers to parents at provider discretion, and initiation of Health interventions by providers as deemed clinically appropriate from their review of the data collected and their knowledge of the participant.
  * Parents will enter home monitoring data daily into the CHAMP App as fitting with their discharge regimen: This may include Feeding, oxygen saturation, heart rate, videos, weight (home scale), or a combination of these.
  Interventions: Device: CHAMP App
- Standard of care control arm (No Intervention): * No proactive monitoring or communication from the research coordinators
  * Follow-up communications from providers to parents at their general healthcare providers discretion, and Initiation of health interventions by providers as deemed clinically appropriate from their review of the data collected and reported by parents via patient portal, phone, and in-person communications and their knowledge of the participant.
  * Parents will be provided a paper log that they will utilize for recording their child's home monitoring data and turn in at the end of the month
  * Parents will write down the home monitoring data fitting with their child's discharge regimen: This may include Feeding, oxygen saturation, heart rate, videos, weight (home scale), or a combination of these.
  * Optional: Parents can utilize the App if they allocate to Arm 2 (Paper) at first, with a combined weekly check-in with the research coordinators. The parents will get a chance to fill out SUS after month of use

INTERVENTIONS:
Device: CHAMP App — CHAMP® App is a proprietary, downloadable, mobile Software Application and software platform designed and developed by the Children's Mercy Hospital of Kansas City (CMH), that permits parents and caregivers to transmit to the care team data to permit remote monitoring of the patient's condition. The parent or caregiver enters into the CHAMP App data including vital signs, intake and output, video, and images of patients (collectively, "CHAMP® Data"), which operates on computers, mobile devices, and handheld computers. The CHAMP® App is intended to be used in the clinical care of pediatric patients in the home setting that are followed by specialty health care teams to improve patient self-management through the use of asynchronous data. Videos and data related to the patient are entered by the parent and sent electronically to the Clinical Care Team as recommended by the clinical team.
  Arms: Proactive Nursing Care model using a mobile application and software platform

SUMMARY:
This is a single-site, stratified grouping parallel- randomized control trial design comparing 30-day all-cause readmission rates and parent experience with two groups of pediatric participants.

DETAILED DESCRIPTION:
This proposal's overall objective is to evaluate the effectiveness of an enterprise-level outpatient nursing care model with an asynchronous mobile health platform for parents of children with medical complexity (CMC) age 0-3 years to communicate with their child's healthcare team via remote patient monitoring (RPM).

The researchers will evaluate the efficacy of a proactive nursing care model on 30-day readmissions (Aim 1), parental experience and managing their child's care at home (Aim 2), and healthcare team engagement frequency with a proactive outpatient nursing care model necessary to achieve adoption into outpatient models of care (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Age 0-3 years 11 months with a parent/Legally authorized representative
* Children with complex medical conditions with medical technologies (feeding, oxygen saturation monitor, and/or oxygen equipment) prescribed by the inpatient care team,
* Discharging to a home setting with parents/legally authorized representatives (LAR's) who can read primarily English, Spanish, Somali, Burmese, Korean, Chinese-Simplified, German, French, Filipino, Arabic, and Vietnamese.
* Availability to download a mobile application onto a parent/LAR-owned device

Additionally, adult participants will also be included and grouped as follows:

Adult Group 1: Parents/Legally authorized representatives of pediatric subject as part of a dyad.

Adult Group 2: Healthcare team users at Children's Mercy Kansas City.

Exclusion Criteria:

* Inability to be discharged to care in the home setting.
* Those not meeting the above inclusion criteria.
* We will exclude a child who is followed solely by the Cardiac High Acuity Monitoring Program Heart Center outpatient team as randomization for this patient population would impact the study design (NCT0603439)
* Those children with PICC lines as their only medical technology.

Equitable Selection: Parent/LAR that do not speak or read one of the 11 languages available in the CHAMP application will be excluded due to potential translation limits of the app.

Healthcare team users: Non-Employees of Children's Mercy.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
All Cause Readmission | 30 days
  During the time period- 30 days after nearest discharge from study enrollment- Any Inpatient or observation encounters to a hospital setting

SECONDARY OUTCOMES:
Home Monitoring Data Adherence | 30 days
  From study enrollment to 30 days after discharge- Remote health monitoring adherence (both arms) to daily data entry
Length of Readmission | 30 days
  Time measured in days of hospital readmission from admission to discharge, Any time of readmission during 30-day monitoring period
Parental Experience | 30 days
  At enrollment and 30 days after discharge: Parental Experience of discharge home after a hospitalization measured by the PACT-M tool at two-time points (enrollment at initial discharge and at 30 days). Along with the data for Aim 1, for the PACT-M tool 35. The PACT-M tool is a 9 item, reliable, validated tool with 5-point Likert answers (Appendix) (Strongly disagree to Agree Strongly). System usability survey questions will also be utilized for Arm 1 CHAMP App participants.
Initiation Adherence | 30 days
  First day of data documentation after discharge
Discontinuation Adherence | 30 days
  Last day of data documentation after discharge before end of study period

OTHER OUTCOMES:
Healthcare Team Engagement | 30 days
  Healthcare team engagement frequency with proactive outpatient nursing care model necessary to achieve adoption into outpatient models of care

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erickson, PhD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will make the data dictionary available on request

REFERENCES:
- [Background] Hall M, Berry JG, Hall M, Goodwin EJ, Margaret Wright S, Bettenhausen J, Colvin JD. Changes in hospitalization populations by level of complexity at children's hospitals. J Hosp Med. 2024 May;19(5):399-402. doi: 10.1002/jhm.13292. Epub 2024 Feb 10. PMID 38340352
- [Background] Shirali G, Erickson L, Apperson J, Goggin K, Williams D, Reid K, Bradley-Ewing A, Tucker D, Bingler M, Spertus J, Rabbitt L, Stroup R. Harnessing Teams and Technology to Improve Outcomes in Infants With Single Ventricle. Circ Cardiovasc Qual Outcomes. 2016 May;9(3):303-11. doi: 10.1161/CIRCOUTCOMES.115.002452. Epub 2016 May 10. PMID 27166202
- [Background] Elliott M, Erickson L, Russell CL, Chrisman M, Gross Toalson J, Emerson A. Defining a new normal: A qualitative exploration of the parent experience during the single ventricle congenital heart disease interstage period. J Adv Nurs. 2021 May;77(5):2437-2446. doi: 10.1111/jan.14785. Epub 2021 Feb 16. PMID 33591609